CLINICAL TRIAL: NCT04211857
Title: A Retro-prospective Follow-up Study of the Safety and Performance of the Round XTENDOBUTTON™ Fixation Device Post Knee Repair in Australian Centres
Brief Title: Retro-prospective Study of Safety & Performance of Round XTENDOBUTTON™ Fixation Device Post Knee Repair
Acronym: XTENDOBUTTON
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: XTENDO.PMCF.2018.12
Record Dates: First submitted 2019-12-23; First posted 2019-12-26 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Knee Reconstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Round XTENDOBUTTON Fixation Device used in suture fixation of ligaments and tendons in conjunction with an ULTRABUTTON™ product or ENDOBUTTON™ device. — Round XTENDOBUTTON Fixation Device used in suture fixation of ligaments and tendons in conjunction with an ULTRABUTTON™ product or ENDOBUTTON™ device.

SUMMARY:
The 12 month post-operative study is designed to provide safety and performance data on the Round XTENDOBUTTON™ fixation device after knee repair.

DETAILED DESCRIPTION:
This is a retro-prospective 12 month follow-up study of the safety and performance of the Round XTENDOBUTTON™ fixation device post knee repair in Australian centres.

The Primary Objective is to assess successful fixation with the Round XTENDOBUTTON™ and the Secondary Objective is to generate safety and performance evidence for the Round XTENDOBUTTON™ Device via the collection of functional outcomes, patient reported outcomes and safety data.

Forty subjects will be enrolled; who have had the round XTENDOBUTTON™ Device implanted. To eliminate the potential for selection bias, Investigators will consecutively screen all subjects who have undergone knee/ligament repair/reconstruction using the Round XTENDOBUTTON™ Fixation Device. Subjects meeting the eligibility criteria will be contacted regarding interest in study participation. Screening will be conducted in sequential order based on the date of subjects' knee repair procedure; earliest to latest. Screening efforts must be documented on a screening and enrollment log, on which reasons for exclusion from or denial to participate should be noted A medical chart review will be conducted to identify potential study subjects who have been implanted with the ROUND XTENDOBUTTON™ device at the study site.

1. If a patient is eligible and would like to participate in the study, obtain written informed consent from the subject.----- Do not proceed until consent has been obtained -----
2. Assign the subject a Subject ID number and instruct the subject on treatment procedures
3. Complete Screening and Enrollment Log
4. Obtain demographic information and medical history, including information on all relevant concomitant medications
5. Collect operative information and implant disposition (including review of evidence of implant failure). If a failure has occurred, record details of the cause of failure. Collect x-rays if available.
6. Complete Patient Questionnaires:

   * Lysholm Score
   * Tegner Activity Scale
   * KOOS(Knee Injury and Osteoarthritis Outcome Score) Knee Score
7. If any adverse events, adverse device effects or device deficiencies are observed or reported, they must be recorded
8. Instruct the subject on follow-up procedures, including returning for Visit 2 in 6 months (-14 Days/+31 Days)

Visit 2 - 12 months post -op.

1. Query subject regarding any changes in general health and the use of concomitant medications since the last visit
2. If any adverse events, adverse device effects or device deficiencies are observed or reported, they must be recorded
3. Complete Lysholm Score, Tegner Activity Scale and KOOS Knee Score
4. Collect implant disposition information (including review of evidence of implant failure). If a failure has occurred, record details of the cause of failure. Collect x-rays if available
5. Complete End of Study CRF.

Safety will be evaluated by assessing the frequency and nature of adverse events, serious adverse events and revisions.

ELIGIBILITY:
Inclusion Criteria:

1. Subject received the Round XTENDOBUTTON™ for knee repair, 6 months (-14 Days/+31 Days) prior to enrollment
2. Subject agrees to follow the prospective study visit schedule (as defined in the study protocol and informed consent form) by signing the IRB/IEC approved informed consent form
3. Subject is ≥ 18 years of age or ≤ 60 years of age at the time of surgery.

Exclusion Criteria:

1. Subject is entered in another investigational drug, biologic, or device study
2. Subjects with a medical or physical condition that, in the opinion of the Investigator, would preclude safe subject participation in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Success of the Round XTENDOBUTTON™ Fixation | 6 months
  The fixation success at 6 months post knee operation with the XTENDOBUTTON™ device. The Kaplan-Meier product limit survival estimates will be presented up to 6 months post-op along with the associated 95% confidence intervals. The event of interest will be fixation failure, defined as a revision due to a device failure, by 6 months.

SECONDARY OUTCOMES:
Fixation success of the Round XTENDOBUTTON™ at 12 months post operation | 12 months
  Fixation success of the Round XTENDOBUTTON™ at 12 months post operation. The Kaplan-Meier product limit survival estimates will be presented up to 12 months post-op along with the associated 95% confidence intervals. The event of interest will be fixation failure, defined as a revision due to a device failure, by 12 months.
Lysholm Score | 6 and 12 months
  The Lysholm Scale evaluates the outcomes of knee ligament surgery. The Lysholm Scale currently consists of eight items that measure: pain (25 points), instability (25 points), locking (15 points), swelling (10 points), limp (5 points), stair climbing (10 points), squatting (5 points), and need for support (5 points). The total score is the sum of each response to the eight questions, and may range from 0-100. Higher scores indicate a better outcome with fewer symptoms or disability
Tegner Activity Scale | 6 & 12 months
  The Tegner activity scale was designed as a score of activity level to complement other functional scores for patients with ligamentous injuries. The Tegner activity scale is a numerical scale ranging from 0 to 10. Each value indicates the ability to perform specific activities. An activity level of 10 corresponds to participation in competitive sports, including soccer, football, and rugby at the elite level; an activity level of 6 points corresponds to participation in recreational sports; and an activity level of 0 is assigned if a person is on sick leave or receiving a disability pension because of knee problems. An activity level of 5 to 10 is recorded only if the patient participates in recreational or competitive sports.
KOOS Score (Knee Injury and Osteoarthritis Outcome Score) | 6 & 12 months
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is self administered and assesses five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee related quality of life.
Adverse events for the study duration | 12 months
Radiographic evaluation at 6 months | 6 months
  Radiographic evaluation will be completed if an implant failure has occurred. Radiographic evaluations (if needed to investigate root cause of a device failure) will be summarized at 6 months.
Radiographic evaluation at 12 months | 12 months
  Radiographic evaluation will be completed if an implant failure has occurred. Radiographic evaluations (if needed to investigate root cause of a device failure) will be summarized at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Sam Chia, MBBS, FRACS (Ortho), FAOrthA, Principal Investigator — PORI- Peninsula Orthopedic Research Institute
Locations (1):
- Peninsula Orthapaedics, Frenchs Forest, Australia

IPD SHARING:
Plan to Share IPD: Yes